CLINICAL TRIAL: NCT05126849
Title: Haploidentical Allogeneic Hematopoietic Stem Cell Transplantation With Post-transplant Cyclophosphamide in Patients With Acquired Refractory Aplastic Anemia or in Relapse After Immunosuppression: a Nationwide Phase II Study
Brief Title: Haploidentical Allogeneic Hematopoietic Stem Cell Transplantation With Post-transplant Cyclophosphamide in Patients With Acquired Refractory Aplastic Anemia or in Relapse After Immunosuppression
Acronym: HAPLO-EMPTY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP200004
Record Dates: First submitted 2021-10-15; First posted 2021-11-19 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Refractory Idiopathic Aplastic Anemia; Haploidentical Allogeneic Hematopoietic Stem Cell Transplantation
Keywords: Acquired refractory idiopathic aplastic anemia; Haplo identical hematopoietic stem cell transplantation; Post-transplantation cyclophosphamide
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Haploidentical allogeneic hematopoietic stem cell transplantation. (Experimental): 1. Conditioning regimen Fludarabine (30mg/m2/day i.v: day -6 to day -2), pre-transplant cyclophosphamide (14.5 mg/kg/day i.v: day -6 and day -5), and Total Body Irradiation (2 Gray on day-1)
  2. Stem cell source Bone Marrow
  3. GVHD Prophylaxis Rabbit ATG dosed at 0.5 mg/kg on day -9 and 2 mg/kg on days -8 and -7, Cyclophosphamide 50 mg/Kg/day at D+3 and D+4, Tacrolimus (residual 8-12 microg/L) and mycophenolate (MMF) from D+5. In absence of GvHD, MMF will be stopped at D35 and tacrolimus at day 365.
  4. Prevention of EBV reactivation Rituximab 150mg/m2 intravenously at Day+5 post HSCT, Each infusion of Rituximab will be preceded by administration of anti-pyretic and an antihistaminic, e.g. paracetamol and diphenhydramine.
  Interventions: Other: Allogenic transplantation

INTERVENTIONS:
Other: Allogenic transplantation — 1. Conditioning regimen Fludarabine (30mg/m2/day i.v: day -6 to day -2), pre-transplant cyclophosphamide (14.5 mg/kg/day i.v: day -6 and day -5), and Total Body Irradiation (2 Gray on day-1)
  2. Stem cell source Bone Marrow
  3. GVHD Prophylaxis Rabbit ATG dosed at 0.5 mg/kg on day -9 and 2 mg/kg on days -8 and -7, Cyclophosphamide 50 mg/Kg/day at D+3 and D+4, Tacrolimus (residual 8-12 microg/L) and mycophenolate (MMF) from D+5. In absence of GvHD, MMF will be stopped at D35 and tacrolimus at day 365.
  4. Prevention of EBV reactivation Rituximab 150mg/m2 intravenously at Day+5 post HSCT, Each infusion of Rituximab will be preceded by administration of anti-pyretic and an antihistaminic, e.g. paracetamol and diphenhydramine.

SUMMARY:
Outcomes for patients with severe aplastic anemia (SAA) who are refractory to first-line immunosuppressive therapy (IST) and who lack a matched unrelated donor (MUD) remain poor. Recently, the use of eltrombopag (ELT) has shown blood count improvements in 40% of these patients. However, most refractory patients do not respond to ELT or other second-line treatment and are therefore exposed to life-threatening infections, and bleeding. During the past 2 decades, there has been a significant decrease in infection-related mortality in patients with SAA unresponsive to initial IST but clonal evolution including paroxysmal nocturnal hemoglobinuria (PNH), myelodysplastic syndrome (MDS), and acute myeloid leukemia (AML) still occur in the long-term with a grim prognosis. Overall, the overall survival of such patients with acquired refractory SAA to ELT is about 60-70% at 2 years.

Hematopoietic stem cell transplantation (HSCT) using alternative donor sources (i.e., mismatched unrelated donors, cord blood (CBT), and haplo-identical family donors) may be curative in patients with refractory SAA, despite carrying much higher rates of complications than in transplantations from matched related or unrelated donors. Recently, our group showed that CBT is a valuable curative option for young adults with refractory SAA. However, not all patients have available CB and CBT treatment related mortality is high in adult patients. Haploidentical (haplo) related donor Stem Cell Transplantation (haplo-SCT) have improved dramatically outcomes using T-cell replete grafts with administration of post-transplantation cyclophosphamide (PTCy). Preliminary results in a little number of patients with refractory SAA at Kings college (London, UK) and John Hopkins (Baltimore, USA) seem promising. The investigators retrospectively analyzed data from 36 patients (median age 42 years) transplanted between 2010 and 2017 in Europe on behalf of the SAA working party of the European Blood and Marrow Transplantation group. The 1-year overall survival was about 80% suggesting that this approach might be a valid option in this particular poor clinical situation.

The main objective of this study is to demonstrate a benefit in term of the 2-year overall survival rate from 60% (historical rates in patients with acquired refractory idiopathic aplastic anemia) up to 80% using haplo-SCT with PTCy.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 3 to 35 years old
* Suffering from refractory acquired idiopathic aplastic anemia (at least one course of immunosuppression with anti-thymocyte globulin)
* Absence of geno-identical donor or 10/10 matched donor
* With identification of a haploidentical donor (brother, sister, parents, adult children or cousin)
* Absence of donor specific antibody detected in the patient with a MFI ≥ 1500 (antibodies directed towards the distinct haplotype between donor and recipient)
* With usual criteria for HSCT :

  * ECOG(Eastern Cooperative Oncology Group) ≤ 2
  * No severe and uncontrolled infection
  * Cardiac function compatible with high dose of cyclophosphamide
* Adequate organ function: ASAT(aspartate transaminase) and ALAT (alanine aminotransferase) ≤ 2.5 N (the norm), total bilirubin ≤ 2N, creatinine < 150 μmol/L
* With health insurance coverage
* Contraception methods must be prescribed during all the duration of the research. Women and men of childbearing age must use contraceptive methods within 12 months and 6 months after the last dose of cyclophosphamide, respectively.
* Having signed a written informed consent (2 parents for patients aged less than 18)

Exclusion Criteria :

* With morphologic evidence of clonal evolution (patients with isolated bone marrow cytogenetic abnormalities are also eligible excepted chromosome 7 abnormalities and complex karyotype)
* With uncontrolled infection
* With seropositivity for HIV or HTLV-1 (Human T cell Leukemia) or active hepatitis B or C defined by a positive PCR (polymerase chain reaction) HBV (hepatitis B virus) or HCV (hepatitis C virus) and associated hepatic cytolysis
* Cancer in the last 5 years (except basal cell carcinoma of the skin or "in situ" carcinoma of the cervix)
* Pregnant (βHCG positive) or breast-feeding.
* Who received live attenuated vaccine within 2 months before transplantation and during the research
* Uncontrolled coronary insufficiency, recent myocardial infarction <6 month, current manifestations of heart failure, uncontrolled cardiac rhythm disorders, ventricular ejection fraction <50%
* With heart failure according to NYHA (New York Heart Association) (II or more)
* Preexisting acute hemorrhagic cystitis
* Renal failure with creatinine clearance <30ml / min
* With urinary tract obstruction
* Who receive the following treatments Phenytoin, Pentostatin, inhibitor of adenoside)
* Who have any debilitating medical or psychiatric illness, which preclude understanding the inform consent as well as optimal treatment and follow-up
* Under tutorship or curatorship

Ages: 3 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Estimated)
Dates: Start 2022-01-06 (Actual); Primary Completion 2027-01-06 (Estimated); Study Completion 2027-01-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | at 2 years

SECONDARY OUTCOMES:
Graft failure incidence | at 2 years
Neutrophils engraftment | at day 100
  3 consecutive days with neutrophiles >0.5 G/L
Platelets engraftment | at day 100
  7 consecutive days with platelets >20 G/L
Absolute numbers of neutrophils | at 1 month
Absolute numbers of neutrophils | at 2 months
Absolute numbers of neutrophils | at 3 months
Absolute numbers of neutrophils | at 6 months
Absolute numbers of neutrophils | at 12 months
Absolute numbers of neutrophils | through study completion, an average of 6 months
Absolute numbers of platelets | at 1 month
Absolute numbers of platelets | at 2 months
Absolute numbers of platelets | at 3 months
Absolute numbers of platelets | at 6 months
Absolute numbers of platelets | at 12 months
Absolute numbers of platelets | through study completion, an average of 6 months
Incidence of use of growth factors for poor hematopoietic reconstitution | up to one year
Acute graft-versus-host disease (GvHD) incidence | at 3 months
Chronic graft-versus-host disease (GvHD) incidence | at 24 months
Relapse incidence | at 12 months
Relapse incidence | at 24 months
Progression free survival | at 12 months
Progression free survival | at 24 months
Incidence of cytomegalovirus (CMV) infection | at 12 months
Incidence of Epstein-Barr virus (EBV) infection | at 12 months
Severe infections (CTAE grade 3-4) | at 3 months
Severe infections (CTAE grade 3-4) | at 6 months
Severe infections (CTAE grade 3-4) | at 12 months
Severe infections (CTAE grade 3-4) | at 24 months
Non-relapse mortality | at 24 months
Incidence of cardiac toxicities | at 12 months
Overall survival | at 12 months
Quality of life questionnaire for adults | at 3 months
  Quality of life will be assessed for adult using "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (QLQ) " EORTC QLQ-C30-V3 questionnaire.The QLQ-C30 is composed of both multi-item scales and single-item measures. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of life questionnaire for minors | at 3 months
  Quality of life will be assessed for minor using The Pediatric Quality of Life Inventory™ (PedsQL™) The 36-item PedsQL™ Family Impact Module is a parent-report instrument designed to assess the impact of pediatric chronic health conditions on parents and the family. It includes 6 subscales measuring parents' self-reported functioning. The scale has five Likert response options, 'never', 'almost never', 'sometimes', 'often' and 'almost always' (corresponding to scores of 100, 75, 50, 25 and 0). Higher scores indicate better functioning.
Quality of life questionnaire for adults | at 6 months
  Quality of life will be assessed for adult using "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" EORTC QLQ-C30-V3 questionnaire.The QLQ-C30 is composed of both multi-item scales and single-item measures. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of life questionnaire for minors | at 6 months
  Quality of life will be assessed for minor using The Pediatric Quality of Life Inventory™ (PedsQL™) The 36-item PedsQL™ Family Impact Module is a parent-report instrument designed to assess the impact of pediatric chronic health conditions on parents and the family. It includes 6 subscales measuring parents' self-reported functioning. The scale has five Likert response options, 'never', 'almost never', 'sometimes', 'often' and 'almost always' (corresponding to scores of 100, 75, 50, 25 and 0). Higher scores indicate better functioning.
Quality of life questionnaire for adults | at 12 months
  Quality of life will be assessed for adults using "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" EORTC QLQ-C30-V3 questionnaire.The QLQ-C30 is composed of both multi-item scales and single-item measures. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of life questionnaire for minors | at 12 months
  Quality of life will be assessed for minor using The Pediatric Quality of Life Inventory™ (PedsQL™) The 36-item PedsQL™ Family Impact Module is a parent-report instrument designed to assess the impact of pediatric chronic health conditions on parents and the family. It includes 6 subscales measuring parents' self-reported functioning. The scale has five Likert response options, 'never', 'almost never', 'sometimes', 'often' and 'almost always' (corresponding to scores of 100, 75, 50, 25 and 0). Higher scores indicate better functioning.
Quality of life questionnaire for adults | at 24 months
  Quality of life will be assessed for adult using "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" EORTC QLQ-C30-V3 questionnaire.The QLQ-C30 is composed of both multi-item scales and single-item measures. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of life questionnaire for minors | at 24 months
  Quality of life will be assessed for minor using The Pediatric Quality of Life Inventory™ (PedsQL™) The 36-item PedsQL™ Family Impact Module is a parent-report instrument designed to assess the impact of pediatric chronic health conditions on parents and the family. It includes 6 subscales measuring parents' self-reported functioning. The scale has five Likert response options, 'never', 'almost never', 'sometimes', 'often' and 'almost always' (corresponding to scores of 100, 75, 50, 25 and 0). Higher scores indicate better functioning.
Proportion of patients with a donor chimerism of 90% or more | at 1 months
Proportion of patients with a donor chimerism of 90% or more | at 3 months
Proportion of patients with a donor chimerism of 90% or more | at 6 months
Proportion of patients with a donor chimerism of 90% or more | at 12 months
Proportion of patients with a donor chimerism of 90% or more | at 24 months
Immune reconstitution by analyzing T, B, natural killer (NK), regulatory T cell levels in the peripheral blood | at 3 months
Immune reconstitution by analyzing T, B, natural killer (NK), regulatory T cell levels in the peripheral blood | at 6 months
Immune reconstitution by analyzing T, B, natural killer (NK), regulatory T cell levels in the peripheral blood | at 12 months
Immune reconstitution by analyzing T, B, NK, regulatory T cell levels in the peripheral blood | at 24 months
Ferritin levels | at 3 months
Ferritin levels | at 6 months
Ferritin levels | at 12 months
Ferritin levels | at 24 months

CONTACTS AND LOCATIONS:
Locations (31):
- France (31):
  - CHU Amiens, Amiens
  - CHU Angers, Angers
  - CHU Besancon, Besançon
  - CHU Bordeaux, Bordeaux
  - Hôpital du Haut-Lévêque, Bordeaux
  - CHU Caen, Caen
  - Hopital Percy, Clamart
  - CHU Clermont, Clermont-Ferrand
  - CHU-Estaing_Clermont Ferrand, Clermont-Ferrand
  - Henri Mondor, Créteil
  - CHU Grenoble, Grenoble
  - CHU Lille, Lille
  - CHU Limoges, Limoges
  - CHU Lyon Sud, Lyon
  - IHOP, CHU Lyon, Lyon
  - Hopital La Timone, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - Hopital Necker, Paris
  - Hopital Robert Debré, Paris
  - Hôpital de La Pitié Salpetriere, Paris
  - Hôpital Saint Antoine, Paris
  - Hôpital Saint Louis, Paris
  - CHU Poitiers, Poitiers
  - CHU Rennes, Rennes
  - Crlcc Henri Becquerel Rouen, Rouen
  - ICLN_Saint Priest En Jarez, Saint-Priest-en-Jarez
  - CHRU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided